CLINICAL TRIAL: NCT01311180
Title: A Phase II Double-Blind, Parallel Group, Randomized, Placebo Controlled Clinical Trial of Sensoril® for Patients With Generalized Anxiety Disorder.
Brief Title: A Clinical Trial to Study the Effects of Sensoril® for Patients With Generalized Anxiety Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Natreon, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Natreon-GAD-02-001
Record Dates: First submitted 2011-03-02; First posted 2011-03-09 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2015-04

CONDITIONS: Generalized Anxiety Disorder
MeSH Terms: conditions — Generalized Anxiety Disorder | interventions — Ashwagandha

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Sensoril® (Experimental)
  Interventions: Drug: Sensoril®
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sensoril® — Start with 250 mg po QAM for 7 days and then 250 mg po bid for 7 weeks
  Other Names: Ashwagandha; Withania somnifera
  Arms: Sensoril®
Drug: Placebo — Start with 250 mg po QAM for 7 days and then 250 mg po bid for 7 weeks
  Arms: Placebo

SUMMARY:
Sensoril - Extracts of Withania somnifera (Ashwagandha in Ayurvedic Medicine) have shown potent anti-stress, cortisol lowering, GABAergic, serotonergic and antioxidant properties in animal and human studies. Furthermore, controlled, single site human studies have shown the anxiolytic potential of WS extracts.The present study is a Phase II Double-Blind, Parallel Group, Randomized, Placebo Controlled Clinical Trial of Sensoril® for Patients with Generalized Anxiety Disorder. The primary objectives of this study are to assess the efficacy and safety of Sensoril® for patients with moderate or greater severity of symptoms associated with Generalized Anxiety Disorder.

The Primary Efficacy endpoint in this study will be determined by a statistically significantly greater improvement from baseline to endpoint in total Hamilton Anxiety Scale scores in the Sensoril® treated group versus those receiving placebo.

The secondary endpoints in this study will assess if Sensoril® treatment rather than placebo results in:

1. Greater response rates (≥ 50% improvement in HAM-A total scores from baseline to last value)
2. Greater remission rates (HAM-A total scores ≤ 7) at week 8
3. Greater improvement from baseline to week 8 in HAM -A psychic and somatic anxiety cluster scores.
4. Greater improvements on CGI - severity scores from baseline to last value.
5. A higher percentage of subjects rated as "much improved" or "very much improved" on the CGI - Improvement subscale at the last value.
6. Serum cortisol and DHEA-S levels will be assessed between the two treatment groups. These biomarkers are indices of stress and it is hypothesized that improvement in levels of these stress indices will favor the Sensoril® treated group.

Exploratory Endpoint

1. Patient reported outcomes for sleep and calmness will be assessed between the two treatments.

Safety Endpoint

The safety endpoints will be determined by assessments of adverse and serious adverse events, physical examination, vital signs, EKG, and clinical laboratory measures. Clinical measures with laboratory defined reference ranges and vital signs will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Adult men and women between the ages of 18 and 65 years (who have completed their 18th birthday but have not completed their 66th birthday) with a Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV TR, APA, 2000) diagnosis of GAD - Generalized Anxiety Disorder.
* Hamilton Anxiety Rating Scale (HAM-A) total score ≥ 20 at the screening and randomization visits.
* HAM-A Item 1 (anxious mood) ≥ 2 at the screening and randomization visits.
* HAM-A Item 2 (tension) ≥ 2 at the screening and randomization visits.
* Montgomery-Asberg Depression Rating Scale (MADRS) total score ≤ 12, with MADRS items #1 and #2 "apparent sadness" and "reported sadness" ≤ 2 at the screening and randomization visits.
* Clinical Global Impression-Severity of Illness (CGI-S) score ≥ 4 at the screening and randomization visits.
* Written Informed Consent present prior to conduct of any study related procedures

Exclusion Criteria:

* Any DSM-IV-TR Axis I disorder other than GAD within 6 months prior to the screening visit.
* Any DSM-IV-TR Axis II disorder that is likely to interfere with the patient's ability to participate in the study.
* Current serious suicidal or homicidal risk, MADRS Item 10 (suicidal thoughts) score > 1, at the screening or randomization visit or a suicide attempt in the 6 months prior to screening.
* Substance or alcohol dependence within 6 months prior to screening. (except Nicotine and/or caffeine)
* Clinically significant deviation from the reference range in clinical laboratory test results during the screening phase and prior to randomization.
* Women who test positive for pregnancy at the screening visit or women who are breast feeding at the screening visit.
* Any thyroid laboratory measures that are considered clinically significant during the screening phase.
* Current (or within past 2 months prior to screening) use of any extract of Withania Somnifera.
* Any known allergy to Withania Somnifera extracts.
* Current (or within the past 2 months prior to screening) over the counter use of herbal extracts such as Ginkgo Biloba, St. John's Wort, Omega-3.
* Specific Concomitant medicines (a table will specify "allowed" and "disallowed" medicines). [Appendix 13]
* Currently (or within the past 2 months prior to screening) receiving any psychotropic medicines (e.g. Anti-anxiety drugs or anti-depressants, or anti-psychotic agents or mood stabilizers).
* Currently (or within the past 2 months prior to screening) receiving any investigational drugs or medical devices.
* Currently (or within the past 2 months prior to screening) undertaking psychotherapy for anxiety or depression.
* Any serious acute or chronic medical condition that in the judgment of the investigator would make it inappropriate for the subject to participate in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2011-03; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Change in the Hamilton Anxiety Rating Scale (HAM-A) total score | 8 weeks
  Mean change from Visit 2 (Baseline) to Visit 7 or Early Termination Visit in HAM-A Total Score.

SECONDARY OUTCOMES:
Change in the Montgomery Asberg Depression Rating Scale (MADRS) total score | 8 weeks
  Mean change from Visit 2 (Baseline) to Visit 7 or Early Termination Visit in MADRS Total Score
Change in the Clinical Global Impression Scales (CGI) for Severity scores. | 8 weeks
  Mean change from Visit 2 (Baseline) to Visit 7 or Early Termination Visit in CGI-Severity Score

CONTACTS AND LOCATIONS:
Locations (7):
- India (7):
  - Asha Hospital, Hyderabad, Andhra Pradesh
  - Sheth V S General Hospital, Ahmedabad, Gujurat
  - Spandana Nursing Home, Bangalore, Karnataka
  - JSS Medical College Hospital, Mysore, Karnataka
  - Sridhar Neuro Psychiatric Center, Shimoga, Karnataka
  - Poona Hospital & Research Centre, Pune, Maharashtra
  - Manobal Medical Research Centre, Lucknow, Uttar Pradesh